CLINICAL TRIAL: NCT03235531
Title: Prospective Assessment of Valproate on Ethanol Withdrawal
Brief Title: Assessment of Valproate on Ethanol Withdrawal
Acronym: PAVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Audis Bethea, Pharm.D., Clinical Pharmacy Specialist, Clinical Research Scientist, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-336
Record Dates: First submitted 2017-07-14; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Alcohol Dependence; Alcohol Withdrawal Syndrome; Trauma; Heavy Drinking; Alcohol Use Disorder
Keywords: alcohol withdrawal syndrome; trauma; alcohol use disorder; alcohol; lorazepam; benzodiazepine; valproate
MeSH Terms: conditions — Alcoholism; Wounds and Injuries | interventions — Valproic Acid; Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CIWA Protocol/BZD and Valproate (Experimental): 1. Interventions to decrease symptoms of AWS will be made based on the CIWA tool.
     * CIWA Score 9-14: 1 mg IV push lorazepam
     * CIWA Score >15: 2 mg IV push lorazepam
  2. Patients who have a known history of alcohol withdrawal seizures or who have received greater than 4 mg IV lorazepam per CIWA protocol will be placed on a scheduled lorazepam regimen, 1 mg every 6 hours. The primary managing service may increase the scheduled lorazepam regimen above 1mg every 6 hours if needed to control withdrawal symptoms. Scheduled lorazepam will be discontinued or de-escalated following a 24-hour period in which no additional lorazepam was received per CIWA protocol.
  3. The treatment group will also receive scheduled valproate (VPA), 15 mg/kg divided over 4 doses, rounded up to the nearest increment of 50mg (i.e. a 70 kg person would be administered 300 mg IV VPA every 6 hours) for 96 hours.
  Interventions: Drug: Valproate; Drug: Lorazepam
- CIWA Protocol Only (Active Comparator): 1. Interventions to decrease symptoms of AWS will be made based on the CIWA tool
     * CIWA Score 9-14: 1 mg IV push lorazepam
     * CIWA Score >15: 2 mg IV push lorazepam
  2. Patients who have a known history of alcohol withdrawal seizures or who have received greater than 4 mg IV lorazepam per CIWA protocol will be placed on a scheduled lorazepam regimen, 1 mg every 6 hours. The primary managing service may increase the scheduled lorazepam regimen above 1mg every 6 hours if needed to control withdrawal symptoms. Scheduled lorazepam will be discontinued or de-escalated following a 24-hour period in which no additional lorazepam was received per CIWA protocol.
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Valproate — Valproate is an anti-epileptic medication that can influence the chemical changes in the brain that result from alcohol withdrawal syndrome (AWS) via three mechanisms of action: (1) an increase in GABA activity, (2) inhibition of glutamate binding to NMDA, and (3) restoration of the balance between dopamine and acetylcholine activity. VPA may be effective in the prevention of AWS, and could serve as efficacious adjuvant to traditional benzodiazepine (BZD) therapy for AWS, both decreasing symptoms of AWS and decreasing the use of BZDs.
  Arms: CIWA Protocol/BZD and Valproate
Drug: Lorazepam — Lorazepam is a benzodiazepine used to treat symptoms of AWS. Standard of care at CAMC is monitoring by CIWA tool and administration of lorazepam according to CIWA score.

SUMMARY:
Alcohol use disorder, or heavy drinking, is commonly seen in patients who present to trauma centers. These patients are at risk for Alcohol Withdrawal Syndrome (AWS), which is collection of symptoms that can range from anxiety and restlessness to seizures, delirium and even death. The Clinical Institute Withdrawal Assessment (CIWA) tool is routinely used to assess alcohol withdrawal symptoms. Benzodiazepines (BZD) are commonly administered to trauma patients who exhibit symptoms of AWS based on the CIWA scoring system. Although these medications have proven efficacy, they can also have negative side effects which may affect recovery. Valprate (VPA) is a medication which may have efficacy in management of AWS symptoms, thus ameliorating or preventing the need for BZD administration. This trial will study the effectiveness of VPA in the prevention of AWS symptoms by comparing the amount of BZD use in trauma patients who receive BZD treatment as indicated by CIWA scores with patients who receive prophylactic VPA therapy in addition to BZD as indicated by CIWA scores.

DETAILED DESCRIPTION:
Alcohol use disorder is a common comorbidity among trauma patients. This pre-existing condition is associated with Alcohol Withdrawal Syndrome (AWS) and frequently complicates the management of this patient population. Current treatment and/or prevention of AWS includes the administration of sedatives (benzodiazepines [BZD]) in response to the manifestation AWS symptoms. This manifestation is indicated by monitoring patients using the Clinical Institute Withdrawal Assessment (CIWA) tool. Benzodiazepines elicit an effect on AWS via mediation of the inhibitory neurotransmitter gamma-aminobutyric acid (GABA). Benzodiazepines, however, have the potential to promote multiple negative effects in the acute care setting, including increased incidence of delirium, hospital stay, mortality, and the potential for decreased long-term cognitive function. The antiepileptic medication valproate (VPA) also has GABA activity in the brain, but may be less likely to promote the negative effects associated with BZDs. Currently, previous experience with this agent for the prevention of AWS is limited to two small studies. In these studies VPA was shown to decrease symptoms of AWS as indicated by patients' CIWA scores. Therefore, VPA could serve as an efficacious adjuvant therapy for the prevention of AWS. The aim of this study is to determine whether VPA will decrease the use of BZD in patients who are receiving symptom-based preventative therapy via CIWA monitoring. The hypothesis is that VPA will decrease the utilization of symptom-based lorazepam administration in patients who are determined to be at risk of alcohol withdrawal due to routine consumption of alcohol.

The purpose of this study is to determine if prophylactic VPA for the prevention of alcohol withdrawal syndrome can decrease symptom-triggered use of benzodiazepines in patients monitored for alcohol withdrawal syndrome with the CIWA.

The Primary objective of this study is to determine if prophylactic VPA acid is associated with decreased lorazepam use in patients monitored for alcohol withdrawal syndrome with the CIWA.

Secondary objectives are:

To evaluate the difference between comparator arms with respect to:

* CIWA scores between patients with and without VPA prophylaxis
* Hospital and Intensive Care Unit (ICU) length of stay
* In-hospital mortality
* VPA acid associated side effects (e.g. thrombocytopenia, transaminitis, pancreatitis)

This will be single-center prospective, randomized study, enrolling trauma patients with a history of alcohol consumption admitted to a Level 1 trauma center. Patients included in this study will receive standard therapies for AWS practiced at study institution which include monitoring of withdrawal symptoms and the administration of BZDs (lorazepam) based on CIWA monitoring.

Following informed consent, patients will be randomized to receive CIWA protocol monitoring/BZD or CIWA protocol monitoring/BZD and VPA. Therefore, patients that meet the inclusion criteria will be separated into two study groups to compare outcomes:

1. Treatment Group: Patients treated with CIWA protocol/BZD and VPA
2. Control Group: Patients treated with CIWA protocol/BZD only.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Trauma Services
* Heavy drinkers based on social history

  * Men <65 years: > 4 drinks per day or 14 per week
  * Women: > 3 drinks per day or 7 drinks per week
  * All adults >65 years: > 3 drinks per day or 7 drinks per week
* Moderate or severe alcohol use disorder based on social history and DSM-5 criteria

  * Moderate: Presence of 4-5 symptoms based on social history
  * Severe: Presence of 6 symptoms based on social history

Exclusion Criteria:

* Intubated patients
* Glasgow Coma Score <8
* Grade IV liver laceration or greater
* Child-Pugh Class B or greater, history of cirrhosis, or cirrhosis identified by radiographic imaging upon admission
* Transaminase (AST/ALT) elevation of ≥ 2x normal
* Anticipated admission less than 72 hours
* Levetiracetam administration for seizure prophylaxis secondary to a traumatic brain injury
* Patient with VPA as home medication
* Known allergy to VPA
* Patients with pre-existing blood dyscrasias, i.e. thrombocytopenia (platelet count < 50,000, etc)
* Inability to obtain social history from patient, surrogate, family member or an individual deemed to be knowledgeable about the patient's social history
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2017-07-11 (Actual); Primary Completion 2019-07-11 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Lorazepam use in patient monitored with CIWA | Time between CIWA initiation and discontinuation for up to 3 weeks
  Amount of lorazepam administration in response to CIWA score

SECONDARY OUTCOMES:
CIWA score | During patient hospital stay for up to 6 months
  CIWA is a ten item scale used in the assessment and management of alcohol withdrawal.
Hospital Length of Stay | During patient hospital stay for up to 6 months
  Date of admission to date of discharge from the hospital
Intensive Care Unit Length of Stay | During patient Intensive Care Unit stay for up to 6 months
  Date of admission to date of discharge from the Intensive Care Unit
In-hospital Mortality | During patient hospital stay for up to 6 months
  Number of deaths
Valproate associated side effects | During patient hospital stay for up to 6 months
  Known side effects associated with valproate use, such as thrombocytopenia, transaminitis, pancreatitis, and hyperammonemia

CONTACTS AND LOCATIONS:
Overall Officials: Audis Bethea, PharmD, BCPS, Principal Investigator — Charleston Area Medical Center Health System
Locations (2):
- United States (2):
  - Charleston Area Medical Center, General Hospital, Level 1 Trauma Center, Charleston, West Virginia
  - Charleston Area Medical Center, Charleston, West Virginia

REFERENCES:
- [Background] Eastes LE. Alcohol withdrawal syndrome in trauma patients: a review. J Emerg Nurs. 2010 Sep;36(5):507-9. doi: 10.1016/j.jen.2010.05.011. Epub 2010 Aug 5. No abstract available. PMID 20837230
- [Background] Craft PP, Foil MB, Cunningham PR, Patselas PC, Long-Snyder BM, Collier MS. Intravenous ethanol for alcohol detoxification in trauma patients. South Med J. 1994 Jan;87(1):47-54. doi: 10.1097/00007611-199401000-00011. PMID 8284718
- [Background] Makic MB. Alcohol Withdrawal Syndrome. J Perianesth Nurs. 2017 Apr;32(2):140-141. doi: 10.1016/j.jopan.2017.01.007. No abstract available. PMID 28343640
- [Background] Foy A, Kay J. The incidence of alcohol-related problems and the risk of alcohol withdrawal in a general hospital population. Drug Alcohol Rev. 1995;14(1):49-54. doi: 10.1080/09595239500185051. PMID 16203295
- [Background] Spies C, Tonnesen H, Andreasson S, Helander A, Conigrave K. Perioperative morbidity and mortality in chronic alcoholic patients. Alcohol Clin Exp Res. 2001 May;25(5 Suppl ISBRA):164S-170S. doi: 10.1097/00000374-200105051-00028. PMID 11391067
- [Background] Tsai G, Gastfriend DR, Coyle JT. The glutamatergic basis of human alcoholism. Am J Psychiatry. 1995 Mar;152(3):332-40. doi: 10.1176/ajp.152.3.332. PMID 7864257
- [Background] Tsai G, Coyle JT. The role of glutamatergic neurotransmission in the pathophysiology of alcoholism. Annu Rev Med. 1998;49:173-84. doi: 10.1146/annurev.med.49.1.173. PMID 9509257
- [Background] McKeon A, Frye MA, Delanty N. The alcohol withdrawal syndrome. J Neurol Neurosurg Psychiatry. 2008 Aug;79(8):854-62. doi: 10.1136/jnnp.2007.128322. Epub 2007 Nov 6. PMID 17986499
- [Background] Amato L, Minozzi S, Davoli M. Efficacy and safety of pharmacological interventions for the treatment of the Alcohol Withdrawal Syndrome. Cochrane Database Syst Rev. 2011 Jun 15;2011(6):CD008537. doi: 10.1002/14651858.CD008537.pub2. PMID 21678378
- [Background] Kosten TR, O'Connor PG. Management of drug and alcohol withdrawal. N Engl J Med. 2003 May 1;348(18):1786-95. doi: 10.1056/NEJMra020617. No abstract available. PMID 12724485
- [Background] Maldonado JR. Delirium in the acute care setting: characteristics, diagnosis and treatment. Crit Care Clin. 2008 Oct;24(4):657-722, vii. doi: 10.1016/j.ccc.2008.05.008. PMID 18929939
- [Background] Clegg A, Young JB. Which medications to avoid in people at risk of delirium: a systematic review. Age Ageing. 2011 Jan;40(1):23-9. doi: 10.1093/ageing/afq140. Epub 2010 Nov 9. PMID 21068014
- [Background] Girard TD, Pandharipande PP, Ely EW. Delirium in the intensive care unit. Crit Care. 2008;12 Suppl 3(Suppl 3):S3. doi: 10.1186/cc6149. Epub 2008 May 14. PMID 18495054
- [Background] Saitz R, Mayo-Smith MF, Roberts MS, Redmond HA, Bernard DR, Calkins DR. Individualized treatment for alcohol withdrawal. A randomized double-blind controlled trial. JAMA. 1994 Aug 17;272(7):519-23. PMID 8046805
- [Background] Eyer F, Schreckenberg M, Hecht D, Adorjan K, Schuster T, Felgenhauer N, Pfab R, Strubel T, Zilker T. Carbamazepine and valproate as adjuncts in the treatment of alcohol withdrawal syndrome: a retrospective cohort study. Alcohol Alcohol. 2011 Mar-Apr;46(2):177-84. doi: 10.1093/alcalc/agr005. PMID 21339186
- [Background] Reoux JP, Saxon AJ, Malte CA, Baer JS, Sloan KL. Divalproex sodium in alcohol withdrawal: a randomized double-blind placebo-controlled clinical trial. Alcohol Clin Exp Res. 2001 Sep;25(9):1324-9. PMID 11584152
- [Background] Lum E, Gorman SK, Slavik RS. Valproic acid management of acute alcohol withdrawal. Ann Pharmacother. 2006 Mar;40(3):441-8. doi: 10.1345/aph.1G243. Epub 2006 Feb 28. PMID 16507623
- [Background] Sher Y, Miller Cramer AC, Ament A, Lolak S, Maldonado JR. Valproic Acid for Treatment of Hyperactive or Mixed Delirium: Rationale and Literature Review. Psychosomatics. 2015 Nov-Dec;56(6):615-25. doi: 10.1016/j.psym.2015.09.008. Epub 2015 Oct 3. PMID 26674479